CLINICAL TRIAL: NCT02708056
Title: Sugammadex Given for the Reversal of Deep Rocuronium Induced Neuromuscular Blockade Under Sevoflurane Anesthesia in Infants: A Retrospective Study
Brief Title: Sugammadex Given for the Reversal of Rocuronium Induced Neuromuscular Blockade Under Sevoflurane Anesthesia in Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ozlem Ozmete, Medical Doctor, Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA 16-67
Record Dates: First submitted 2016-02-25; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Brain Cancer
Keywords: Sugammadex; Rocuronium; Infant patients
MeSH Terms: conditions — Brain Neoplasms | interventions — Sugammadex

ARMS (1):
- Sugammadex, Bridion (Other): Drug were given intravenously by a anesthesiologist at the end of surgery
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex
  Other Names: Bridion

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of sugammadex in reversing profound neuromuscular block induced by rocuronium in infant patients

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 1-12 month,
* ASA physical status 1-3 who underwent elective brain cancer surgery during general anesthesia were included in the study

Exclusion Criteria:

* younger than 1month or older than 12 months.
* hepatic or renal failure
* A history of allergy to study medication

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The efficacy of sugammadex were assessed by using Train of four (TOF) | 1 year